CLINICAL TRIAL: NCT06176859
Title: Delivery Optimization for Pre-Exposure Prophylaxis (DO PrEP) Study: A Prospective, Interventional, Randomized Study of Community-based PrEP Initiation, Delivery, and Monitoring in South Africa
Brief Title: Delivery Optimization for Pre-Exposure Prophylaxis (DO PrEP) Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, MBChB, MSc, DPhil., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P003023
Record Dates: First submitted 2023-04-22; First posted 2023-12-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV; Human Immunodeficiency Virus; ART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective, interventional, and randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Home-based PrEP (Experimental): In the home-based PrEP arm, participants will complete the HIV self-test at home with support received through telemedicine or over the phone. Confirmation of HIV test result will be shared with the provider through a photograph of the test. PrEP refills will be delivered to participants at home by courier.
  Interventions: Other: HIV PrEP Delivery
- Community-based PrEP (Active Comparator): In the community-based PrEP arm, participants will be tested using rapid diagnostic tests (RDT) in person (at a community venue) or through telemedicine (at a community venue) where they will be linked by counsellor telephonically to nurse or clinician. PrEP refills will be collected by participants at a community venue.
  Interventions: Other: HIV PrEP Delivery

INTERVENTIONS:
Other: HIV PrEP Delivery — To test an end-to-end decentralized delivery service for pre-exposure prophylaxis (PrEP) to safely increase PrEP access and use among priority populations in South Africa.

SUMMARY:
The overall goal is to determine whether an end-to-end decentralized delivery service for PrEP is more effective, safe, acceptable, and cost-effective than facility-based PrEP delivery.

DETAILED DESCRIPTION:
Optimizing pre-exposure prophylaxis (PrEP) delivery with a focus on priority populations is critical to realize the enormous potential of PrEP for HIV prevention. HIV incidence remains relentlessly high among young women and sexual minority men and primary prevention is critical to achieving control of the HIV epidemic. With effective and persistent use, oral pre-exposure prophylaxis (PrEP) for HIV prevents 75%-100% of HIV cases among cisgender women and men, gay and bisexual men, and transgender women. Despite the high efficacy, uptake throughout the PrEP prevention cascade remains low.

South Africa is expanding PrEP provision but requires evidence-based strategies on how to achieve access, effective use, and persistence. The current clinic-based requirement of PrEP to persons at risk for HIV acquisition requires that clients self-identify their exposure to HIV and visit the clinic regularly for initiation, monitoring and refills. Barriers to PrEP access include clinic level factors (i.e. staff training, brief visits) and individual level factors including logistics such as transportation for clinic visits. The priority is to determine how to deliver PrEP in a scalable way and achieve high PrEP access and effective, persistent use.

PrEP is a highly efficacious HIV prevention strategy but requires effective strategies that streamline delivery and engage users for scale-up. Community-based strategies for HIV testing, ART initiation, and monitoring successfully reach people living with HIV for treatment and have made marked improvements to viral suppression.

This protocol describes a randomized clinical study to test an end-to-end decentralized delivery service for PrEP. It aims to safely increase PrEP access and use among priority populations in South Africa. Participants will include 16-30 year old HIV negative women and sexual minority men at high risk for acquiring HIV. As a critical component of decentralized delivery, we will also evaluate the safety and efficacy of HIV self-testing compared to rapid diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years - 30 years old,
* Self-report living without HIV or unknown status.
* Persons who have been sexually active within the last 3 months
* Interested in the use of PrEP for HIV prevention.
* Able and willing to provide informed consent for study procedures.
* Access to a cellphone for study related communication
* Reside in the study community for the duration of follow-up.

Exclusion Criteria:

* HIV infection based on negative HIV rapid tests
* Clinically ineligible for PrEP
* The participant doesn't reside in the study community for the duration of follow-up

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2500 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is uptake of Pre-exposure prophylaxis of HIV (PrEP) . | 36 Months
  The proportion of study participants who effectively accessed PrEP and continued use over a 12-month period.

SECONDARY OUTCOMES:
The efficacy of rapid HIV testing kits in diagnosing HIV for PrEP initiation. | 36 Months
  To compare the safety and efficacy of HIV self-testing (HIVST) to rapid diagnostic tests (RDT) by comparing the sensitivity and specificity of each diagnostic test.
Persistent use of PrEP over a 12-month period. | 36 Months
  The proportion of study participants in the home-monitored arm who accessed and effectively/persistently used PrEP over a 12-month period compared to the community-monitored arm.
Cost effectiveness per HIV incident averted. | 36 Months
  Estimate the incremental cost-per-person receiving community-based PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Zaynab Essack, PhD, Principal Investigator — Human Sciences Research Council of South Africa
Locations (1):
- Human Sciences Research Council, Durban, KwaZulu-Natal, South Africa